CLINICAL TRIAL: NCT05522140
Title: Testing the Effectiveness of a Nature-based Social Intervention on Loneliness Among Lonely Adults in Prague - a Randomized Controlled Trial
Brief Title: Testing a Nature-based Socila Intevention on Loneliness: the RECETAS-PRG Trial
Acronym: RECETAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vladimíra Dostálová (Other)
Collaborators: Barcelona Institute for Global Health (Other)
Responsible Party: Sponsor-Investigator, Vladimíra Dostálová, Senior researcher, Charles University, Czech Republic
Organization: Charles University, Czech Republic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 945095 PRG
Record Dates: First submitted 2022-08-25; First posted 2022-08-30 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Loneliness
Keywords: social prescribing; social intervention; nature-based activities; mental health; wellbeing; prevention; nature-based therapy; complex intervention; community-based; urban health; loneliness
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): The intervention arm will undergo following steps:
  1. Groups of 5-15 persons, who lives in Prague. Two trained facilitators support the group dynamics forstering empowerment.
  2. Each participant will undergo an individual session with the facilitator(s) aimed at building relationships and trust, and getting to know the expectations and characteristics of the participants.
  3. 9 group activities with the aim to promote accessibility and engagement with the nature and outdoor activities available in their town. Collaborative mapping of nature-based community activities will direct the group to activities they want to approach and test.
  Interventions: Behavioral: Nature-based social intervention (NBIS)
- Control arm (Active Comparator): Participants randomly assigned to the control arm will receive usual care, which is a list of community resources in the city (Prague). Usual care is an appropriate comparison rather than placebo for complex interventions
  Interventions: Behavioral: Usual care + menu with nature based activities

INTERVENTIONS:
Behavioral: Nature-based social intervention (NBIS) — Nature-based social prescribing is a multicomponent, multi-level, behaviorally based complex intervention applaied by facilitators after a specific training. It comprises: a psychosocial component and nature-based activities. The psychosocial component is adapted from the group dynamic of "Circle of Friends" methodolgy focused on loneliness(Jansson A, Pitkälä KH, 2021) adapted to the cultural context of Prague and the target population (partitipants) of adults who lives in Prague. Participants start with an individual session and then meet once a week for two hours for 10 weeks.
  At the first meeting together, participants select the nature-based activities they wish to conduct through a co-created menu.
  Arms: Intervention arm
Behavioral: Usual care + menu with nature based activities — Social prescribing as existing in usual care plus a written menu with the list of nature-based activities in the area.
  Arms: Control arm

SUMMARY:
RECETAS (Re-imagine Environments for Connection and Engagement: Testing Actions for Social Prescribing in Natural Spaces) is an European project (H2020 No 945095) that aims to reduce loneliness by linking lonely pople to nature-based social actvitities through a group-based intervention.

Background: Loneliness is a person's own perception when his/her need for satisfying social contact and relationships is not met. The feeling of loneliness can be experienced even by a person who is surrounded by people. RECETAS aims to design and test nature-based socila itervention (NBSI) that is group-based and includes access to nature as a main component. The testing will be conducted in six different citites: Barcelona, Helsinki, Prague, Marseille, Cuenca in Ecuador and Melbourne. If succesful, this will provide an evidence-based approach for using social prescribing to address loneliness.

Objectives: to assess the effectiveness of a 10-week NBSI on loneliness and health-related quality of life in vulnerable people in the area of Prague suffering from it compared to usual social and health care at post-intervention, and at 6-, and 12-months post-randomization.

A pilot study was conducted from May to June 2022 prior to the start of the study in January 2023. The main aim of the pilot study was to identify barriers and obstacles to conducting the trial itself.

Methods: The study design is a randomized controlled trial (RCT) including a process evaluation based on Medical health Council guidance, a nested qualitative study and a Health Economics evaluation.

Participants will be recruited mainly from primary care settings (health and social), third sector organisations, community groups, and volunteer organisations. A total of 316 participants will be randomly allocated in two arms after the baseline assessment: NBSI tratment and control arms. All of them will be asked to sign the informed consent form.

DETAILED DESCRIPTION:
RECETAS (Re-imagine Environments for Connection and Engagement: Testing Actions for Social Prescribing in Natural Spaces) is project that adresses loneliness and the role of nature-based social prescription (NBSP) to reduce it. This project has received funding from European Union's Horizon research and innovation under grant agreement No 945094. More information at: https://recetasproject.eu/

Background: Loneliness is a person's own perception when his/her need for satisfying social contact and relationships is not met. The feeling of loneliness can be experienced even by a person who is surrounded by people. Loneliness is a modifiable health condition that is potentially dangerous to health and can reduce people's life span. In Europe, 30 million people European adults frequently felt lonely.

Social prescription is a non-medical approach that aims to connect people with the community through social outdoor activities to improve their wellbeing. NBSP is an intervention where nature-based social activities connect people, places and institutions that form strong social networks and connections. Nature-based activities can facilitate a dynamic process and social interactions and can thus contribute to reducing feelings of loneliness. We will design and test nature-based social intervention (NBSI) that is group-based and includes access to nature as a main component. The testing will be conducted in six urban areas: Barcelona, Helsinki, Prague, Cuenca in Ecuador and Melbourne.

Objectives: to assess the effectiveness of a 10-week NBSI on loneliness and health-related quality of life in vulnerable people in the area of Prague suffering from it compared to usual social and health care at post-intervention, and at 6-, and 12-months post-randomization.

A pilot study was conducted from May to June 2022 prior to the start of the study in January 2023. The main aim of the pilot study was to identify barriers and obstacles to conducting the trial itself.

Methods: A randomized controlled trial (RCT) will be used to assess the effect of NBSI on reducing feelings of loneliness. The RCT will use mixed-method approach collecting qunatitative information to assess the the main outcomes and qualitative methods to explore participant's and professional's experiences. ISGlobal coordinates the overall RECETAS project. Charles University leads the implementation of the RECETAS-PRG and is responsible for the recruitment process, intervention, assessment, evaluation, data analysis and qualitative part of the study.

Recruitment will be carried out in cooperation with the Centre of Longevity and Long-Term Care, the Czech Alzheimer's Society, general practitioners and other outpatient specialists, and home care organizations based on a long-term focus on the target group. Participants will be recruited mainly from primary care settings (health and social), third sector organisations, community groups, and volunteer organisations. A total of 316 participants will be randomly allocated in two arm (158 each): NBSP intervention arm and control arm. All of them will be asked to sign the informed consent form.

The intervention is a theory-informed, multicomponent, multi-level, behaviorally based complex intervention that requires a specific trainning to prepare facilitators. The intervention model is adapted from the "Circle of Friends" methodology developed by the University of Helsinky by Pitkälä KH et al. It consists in: a) individualized session with facilitators (one-to-one); b) group-based program (5-15 people) for 9 sessions, one a wiil, including nature-based activities in the area chosen by the participants. Control group participants will recieve usual care, and list of natrure-based activities available ti their area.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give informed consent in Czech
2. Older adults (60+) with a risk of social isolation and loneliness
3. Currently experiencing loneliness according to the screening question "Do you suffer from loneliness?"
4. Willing to undergo study measurement.

Exclusion Criteria:

1. Unable to go outdoors due to poor mobility or severe diseases.
2. Poor hearing or sight in case it prevents them to participate of the group dynamics and activities in the nature.
3. Severe, moderate or mild cognitive decline.
4. Any mental health disorders that might interfere with the group dynamics.
5. Severe disease with poor prognosis < 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
De Jong Gierveld Loneliness Scale 11 item | Post-intervention (10 weeks)
  Change in loneliness. De Jong Gierveld Loneliness Scale (minimum 0 (best) and maximum 11 (worst))
15D instrument of health-related quality of life | Post-intervention (10 weeks)
  Change in health related quality of life. Minimum 0 (worst) and maximum 1 (best). 15D will be used as an index ( 0 to 1) and the changes in various 15 dimensions will also be explored.

SECONDARY OUTCOMES:
Psychological Wellbeing Scale by Routasalo et al. 2009 | From baseline to 3months, 6months, 12 months
  Change in psychological wellbeing.Minimum 0 (worst) and maximum 1 (best).
Clock drawing test | From baseline to 3months, 6months, 12 months
  Change in executive function. Minimum 0 (worst) and maximum 6 (best)
Instrumental Activities of Daily Living Scale | From baseline to 3months, 6months, 12 months
  Change in instrumental activities of daily living. Minimum 0 (worst) and maximum 10 (best)
15D instrument of health-related quality of life | Baseline (before intervention), 6- and 12-months follow up
  Change in health related quality of life. Minimum 0 (worst) and maximum 1 (best). 15D will be used as an index ( 0 to 1) and the changes in various 15 dimensions will also be explored.
De Jong Gierveld Loneliness Scale 11 item | Baseline (before intervention), 6- and 12-months follow up
  Change in loneliness. De Jong Gierveld Loneliness Scale (minimum 0 (best) and maximum 11 (worst))
International Physical Activity Questionnaire | From baseline to 3months, 6months, 12 months
  Change in physical activity. Minimum 1 (worst) and maximum 3 (best)
Geriatric Depression Scale | From baseline to 3months, 6months, 12 months
  Change in depression. Minimum 0 (best) and maximum 15 (worst)
Lubben Social Network Scale | From baseline to 3months, 6months, 12 months
  Change in social network. Minimum 0 (worst) and maximum 5 (best)
EURO-QOL 5D-5L | From baseline to 3months, 6months, 12 months
  Health economic analyses. Cost of health services with EQ5D-5L
ICEpop CAPability mesure for Adults (ICECAP-A) | From baseline to 3months, 6months, 12 months
  Self-reported measure of capability wellbeing for adults
Nature connection index | From baseline to 3months, 6months, 12 months
  Relationship with nature. Min = 1 Max = 7. Higher scores indicating stronger connectedness to nature

CONTACTS AND LOCATIONS:
Overall Officials: Jill S Litt, PhD, Principal Investigator — Barcelona Institute for Global Health
Locations (1):
- Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Litt, J. S., Coll-Planas, L., Sachs, A. L., Rochau, U., Jansson, A., Dostálová, V., … Pitkälä, K. H. (2024). Nature-based social interventions for people experiencing loneliness: the rationale and overview of the RECETAS project. Cities & Health, 8(3), 418-431. https://doi.org/10.1080/23748834.2023.2300207
- [Background] Coll-Planas L, Carbo-Cardena A, Jansson A, Dostalova V, Bartova A, Rautiainen L, Kolster A, Maso-Aguado M, Briones-Buixassa L, Blancafort-Alias S, Roque-Figuls M, Sachs AL, Casajuana C, Siebert U, Rochau U, Puntscher S, Holmerova I, Pitkala KH, Litt JS. Nature-based social interventions to address loneliness among vulnerable populations: a common study protocol for three related randomized controlled trials in Barcelona, Helsinki, and Prague within the RECETAS European project. BMC Public Health. 2024 Jan 13;24(1):172. doi: 10.1186/s12889-023-17547-x. PMID 38218784
- [Background] Vert C, Litt JS, Gascon M, Roque M, Maso-Aguado M, Opacin N, Garcia G, Jansson A, Cattaneo L, Bartova A, Briones-Buixassa L, Carbo A, Rautiainen LJ, Hidalgo L, Sachs A, Domenech S, Blancafort-Alias S, Holmerova I, Pitkala KH, Coll-Planas L. Evaluating the feasibility of "Friends in Nature," a complex nature-based social intervention to address loneliness and quality of life in six cities worldwide. Pilot Feasibility Stud. 2024 Nov 30;10(1):146. doi: 10.1186/s40814-024-01575-4. PMID 39616375
- [Background] Sachs AL, Maso-Aguado M, Bach A, Opacin N, Hill N, Cattaneo L, Coll-Planas L, Johnson K, Hidalgo L, Daher C, Litt J, Bekessy S. Developing a new tool to capture the nature dose to reduce loneliness and improve quality of life. MethodsX. 2024 Sep 19;13:102969. doi: 10.1016/j.mex.2024.102969. eCollection 2024 Dec. PMID 39385940
- [Background] Girdler NM. Air-gun injury to the face. Oral Surg Oral Med Oral Pathol. 1994 Aug;78(2):137. doi: 10.1016/0030-4220(94)90133-3. No abstract available. PMID 7936578
- See also: website of the European Projecte RECETAS — http://recetasproject.eu/